CLINICAL TRIAL: NCT03416218
Title: Prognosis--A Game-Based Intervention to Improve STEM Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB17-1416
Record Dates: First submitted 2018-01-05; First posted 2018-01-31 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: STEM Skills
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Participants enrolled in the study will play Prognosis, a game-based intervention designed to improve STEM skills.
Masking Description: There is only one condition to this study, so no masking will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants enrolled in the study will play Prognosis, the intervention being assessed in this study.
  Interventions: Behavioral: Prognosis

INTERVENTIONS:
Behavioral: Prognosis — Prognosis will be a single-player 2D, digital simulation game and supporting multimedia website. Players are situated as a major official of Hexacago, and tasks them with managing the city's finances, education levels, and health concerns to lower rates of teenage pregnancy and sexually transmitted infections. In the game Prognosis, player dispatches professionals from a variety of fields to different neighborhoods around the city, observing the effects of their resource allocation decisions across multiple systems over many in-game months. The supporting multimedia website will house curriculum and learning tools to support the learning objectives of Prognosis.

SUMMARY:
The purpose of this study is to evaluate a game-based intervention (Prognosis) designed to improve science, technology, engineering, and mathematics (STEM) skills among high school-aged students.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the usability, feasibility, and acceptability of a game-based intervention (Prognosis) designed to improve science, technology, engineering, and mathematics (STEM) skills among high school-aged students. The research questions are as follows:

H1: Students will find Prognosis usable, feasible, and acceptable and recommend continued development and testing of Prognosis.

H2: After playing Prognosis, students will be able to perform basic quantitative data skills such as calculating incidence and prevalence.

H3: After playing Prognosis, students will be able to observe patterns in data at the neighborhood and city level.

H4: After playing Prognosis, students will be able to construct explanations and models describing the organization of systems in the game and how they contribute to health outcomes.

H5: After playing Prognosis, students will be able to formulate and test hypotheses for how to best coordinate various city systems and leverage finite resources to reach their target health goal.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in study site high school
* 9th or 10th grade at time of study

Exclusion Criteria:

* Students not in 9th and 10th grade

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of the game-based intervention Prognosis as assessed by participants | immediately after completing the intervention
  questionnaire
Feasibility of the game-based intervention Prognosis | immediately after completing the intervention
  questionnaire
Usability of the game-based intervention Prognosis | immediately after completing the intervention
  questionnaire

SECONDARY OUTCOMES:
Assessing participants' ability to solve quantitative epidemiological problems | immediately after completing the intervention
  Administered through a survey, questions derived from the Principles of Epidemiology in Public Health Practice, Third Edition, An Introduction to Applied Epidemiology and Biostatistics https://www.cdc.gov/ophss/csels/dsepd/ss1978/lesson1/index.html
Perceived self-efficacy to learn STEM concepts | immediately after completing the intervention
  5 questions asking students about their perceived self-efficacy relating to achieving learning objectives. Developed for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States